CLINICAL TRIAL: NCT06758973
Title: Validity and Reliability of the Turkish Version of the 4-Item Short Form of the PASS
Brief Title: Validity and Reliability of the Turkish Version of the 4-Item Short Form of the Pain Anxiety Symptom Scale
Status: Enrolling by invitation | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-009
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Scale Reliability Validity
Keywords: pain; anxiety; reliability; validity
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group

SUMMARY:
The primary aim of the study was to determine the reliability and validity of the Turkish version of the 4-Item Short Form of the Pain Anxiety Symptom Scale. The secondary aim of the study was to determine the level of pain-related anxiety in individuals with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-65
2. Having pain 4 or more days a week
3. Having weekly pain intensity of 3 or more according to the Numeric Pain Rating Scale
4. Having chronic pain lasting at least 3 months
5. Being able to read and write and having no cognitive problems
6. Individuals who volunteer to participate in the study will be included.

Exclusion Criteria:

1. Having pain limited to headache only

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be implemented at the Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center between the dates after receiving the ethics committee approval. Patients who apply to the Physical Medicine and Rehabilitation Polyclinic with complaints of pain will be examined by a physical therapist. Patients who are diagnosed with chronic pain through physical examination, meet the inclusion criteria and agree to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-07-11 (Estimated)

PRIMARY OUTCOMES:
Pain Anxiety Symptom Scale 4-Item Short Form | 20 weeks

SECONDARY OUTCOMES:
Chronic Pain Admission Form | 20 weeks
Beck Anxiety Inventory | 20 weeks
Visual Analog Scale | 20 weeks
Chronic Pain Acceptance Questionnaire | 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No